CLINICAL TRIAL: NCT05674630
Title: TicIn for the Treatment of coronAry lesioNs With Drug Eluting Balloons
Brief Title: Ticin for the Treatment of Coronary Lesions With Drug Eluting Ballons
Acronym: TITAN-DEB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiocentro Ticino (Other)
Collaborators: University of Bern (Other)
Responsible Party: Principal Investigator, Marco Valgimigli, Coordinating Principal Investigator, Cardiocentro Ticino
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01_TITAN-DEB
Record Dates: First submitted 2022-12-07; First posted 2023-01-06 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Chronic Coronary Syndrome
Keywords: adult; chronic coronary syndrome; percutaneous intervention; significant de novo coronary lesion; FFR≤0.80; iFR≤0.89; long DES (≥30 mm); coronary lesion; drug eluting balloon; drug eluting stent; Magic Touch drug eluting balloon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magic Touch drug eluting balloon based strategy - 6/12 months invasive follow up (Experimental): Patients randomized to DEB-based strategy will receive treatment with DEB (Magic Touch, Concept Medical®) throughout the entire lesion length, followed by final assessment with FFR and IVUS at 6 or 12 months in a randomized fashion.
  Interventions: Device: Magic Touch drug eluting balloon based strategy
- Drug eluting stent based strategy - 6/12 months invasive follow up (Active Comparator): Percutaneous transluminal coronary angioplasty and drug eluting stent implantation according to local standard of care, including optimization techniques (e.g. post-dilatation) which are left at operators' discretion, followed by final assessment with FFR and IVUS at 6 or 12 months in a randomized fashion.
  Interventions: Device: Drug-eluting stent-based strategy

INTERVENTIONS:
Device: Magic Touch drug eluting balloon based strategy — Adult patients with chronic coronary syndrome deemed suitable for percutaneous intervention and significant long de-novo coronary lesion randomized in the experimental arm will receive treatment with drug eluting balloon (Magic Touch®) followed by invasive follow up (FFR and IVUS) at 6 ot 12 months in a randomized fashion.
  Arms: Magic Touch drug eluting balloon based strategy - 6/12 months invasive follow up
Device: Drug-eluting stent-based strategy — Adult patients with chronic coronary syndrome deemed suitable for percutaneous intervention and significant long de-novo coronary lesion randomized in the control arm will receive treatment with drug-eluting stent followed by invasive follow up (FFR and IVUS) at 6 ot 12 months in a randomized fashion.
  Arms: Drug eluting stent based strategy - 6/12 months invasive follow up

SUMMARY:
The goal of this clinical trial is to compare the use of a specific drug eluting balloon (Magic Touch, Concept Medical®) versus standard drug eluting stent based strategies in patients with long coronary lesions.

Participants with chronic coronary disease and long coronary stenosis will be randomly assign to be treated either with Magic Touch balloon or drug eluting stent.

DETAILED DESCRIPTION:
Patients at coronary angiography who are deemed suitable for PCI are assessed for eligibility. Patients fulfilling all inclusion and no exclusion criteria can be consented for trial participation. After successful lesion preparation, defined as residual stenosis less than 30%, TIMI flow 3 and no major (type C) dissection of target lesion, consented patients will be randomized in a 1:1 ratio to a drug eluting balloon(DEB)-based or standard drug eluting stent(DES)-based strategy and further randomized in a 1:1 fashion, stratified based on DEB vs DES, to undergo invasive follow-up at 6 (±30 days) or 12 (±30 days) months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years old) with chronic coronary syndrome deemed suitable for PCI
2. At least one significant de-novo coronary lesion (defined as diameter stenosis > 50% on angiography, with flow limiting features, confirmed with FFR ≤0.80 or iFR ≤0.89 and intended implantation of a long (≥30 mm) DES based on IVUS findings
3. Written informed consent

Exclusion Criteria:

1. Patients referred to the index procedure for an acute coronary syndrome
2. Target lesion involving the left main and/or ostial left coronary artery, ostial left circumflex artery or ostial right coronary artery
3. Severe renal impairment (eGFR<15ml/min/1.73m2) or patient on dialysis treatment
4. Spontaneous coronary artery dissection (SCAD)
5. Contraindications to adenosine administration (e.g. moderate to severe asthma or chronic obstructive pulmonary disease, heart rate <50 beats/min and systolic blood pressure <90 mmHg)
6. Known pregnancy or breast-feeding patients
7. Life expectancy <1 year due to other severe non-cardiac disease
8. Legally incompetent to provide informed consent
9. Participation in another clinical study with an investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Absolute change of FFR values (ΔFFR) | At 6(±30days) or 12(±30 days) months after the index PCI
  Absolute change of fractional flow reserve (FFR) values (ΔFFR) measured at the final assessment immediately after the index PCI and invasive follow-up at 6(±30days) or 12(±30 days) months

SECONDARY OUTCOMES:
QCA parameter (minimal lumen diameter, MLD, mm) before and after the intervention and at follow-up angiography | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Minimal lumen diameter (MLD,mm) before the intervention, immediately after the intervention and at follow-up angiography.
QCA parameter (maximal diameter stenosis, MaxS, percent) before and after the intervention and at follow-up angiography | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Maximal diameter stenosis (MaxS, percent) before the intervention, immediately after the intervention and at follow-up angiography.
QCA parameter (reference vessel diameter, RVD, mm) before and after the intervention and at follow-up angiography | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Reference vessel diameter (RVD, mm) before the intervention, immediately after the intervention and at follow-up angiography.
QCA parameter (lesion length, LL, mm) before and after the intervention and at follow-up angiography. | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Lesion length (LL, mm) before the intervention, immediately after the intervention and at follow-up angiography.
QFR parameters before and after intervention and at follow-up angiography | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Quantitative Flow Ratio (QFR) parameters before the intervention, immediately after the intervention and at follow-up angiography
FFR parameters before and after intervention and at follow-up angiography | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Fractional Flow Reserve (FFR) parameters before the intervention, immediately after the intervention and at follow-up angiography
Minimal lumen diameter (MLD, mm) | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Minimal lumen diameter (MLD, mm) evaluated with intravascular ultrasound (IVUS)
Minimal luminal area (MLA, mm^2) | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Minimal luminal area (MLA, mm^2) evaluated with intravascular ultrasound (IVUS)
Maximal diameter stenosis (MaxS, percent) | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Maximal diameter stenosis (MaxS, percent) evaluated with intravascular ultrasound (IVUS)
Lumen volume (LV, mm^3) | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Lumen volume (LV, mm^3) evaluated with intravascular ultrasound (IVUS)
Vessel volume (VV, mm^3) | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Vessel volume (VV, mm^3) evaluated with intravascular ultrasound (IVUS)
Plaque burden (VV-LV) | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Plaque burden (VV-LV) evaluated with intravascular ultrasound (IVUS)
Late lumen loss (LLL) | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Late lumen loss (LLL) evaluated with intravascular ultrasound (IVUS)
Acute gain | pre procedure and immediately after the procedure
  Variation between pre treatment (T0) and immediately after the treatment (Tf)
Disease progression after index PCI | pre procedure, immediately after the procedure and at 6(±30days) or 12(±30 days) months after the index PCI
  Variation between final result of index PCI (Tf) and procedure at 6(±30days) or 12(±30 days) months after the index PCI (Tc)
Target lesion revascularization (TLR) defined as urgent and non-urgent | 5 years after the index PCI
  Rate of target lesion revascularization (TLR) defined as urgent and non-urgent
Target vessel revascularization (TVR), defined as urgent and non-urgent | 5 years after the index PCI
  Rate of target vessel revascularization (TVR), defined as urgent and non-urgent
Target vessel failure (TVF), defined as cardiac death, target-vessel myocardial infarction, and any target lesion revascularization | 5 years after the index PCI
  Rate of target vessel failure (TVF), defined as cardiac death, target-vessel myocardial infarction, and any target lesion revascularization
The individual components of the composite target vessel failure (TVF) endpoint (defined as cardiac death, target-vessel myocardial infarction and any target lesion revascularization) | 5 years after the index PCI
  Rate of the individual components of the composite target vessel failure (TVF) endpoint (defined as cardiac death, target-vessel myocardial infarction and any target lesion revascularization)
Any myocardial infarction | 5 years after the index PCI
  Rate of any myocardial infarction
Stroke | 5 years after the index PCI
  Rate of stroke
Definite or probable stent thrombosis | 5 years after the index PCI
  Rate of definite or probable stent thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Marco Valgimigli, M.D., Ph.D, Principal Investigator — Cardiocentro Ticino Institute, Ente Ospedaliero Cantonale, Lugano,
Locations (1):
- Marco Valgimigli, Lugano, Switzerland